CLINICAL TRIAL: NCT03515330
Title: A Pilot Study of Mobile Directly Observed Therapy (mDOT) for Immunosuppressant Adherence in Adult Liver Transplant Recipients
Brief Title: A Pilot Study of mDOT for Immunosuppressant Adherence in Adult Liver Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Merged IRB study created
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00173000
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Medication Adherence; Liver Transplant
Keywords: mHealth; liver transplantation; medication adherence; video directly observed therapy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a single center, prospective, randomized control trial with two arms. Participants in the intervention arm will use the mHealth app to manage and track their immunosuppression medical regimen post-transplant, and participants in the control arm will receive the current standard of follow-up care post-transplant.
Who Masked: Outcomes Assessor
Masking Description: Patients will be aware of which arm they are randomized to; thus, the study will not be blinded to practitioners or patients. However, study personnel performing data analysis will receive de-identified data that does not explicitly describe which group is intervention and which is control, but simply the code without a key. Only the PI and necessary personnel performing data extraction will have the key for the code to minimize bias in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants in the control arm will be instructed to take their immunosuppressant medications as prescribed and attend required follow-up as is standard of care, and will not receive the mHealth application.
- mHealth Intervention (Experimental): Participants in the intervention arm will receive the mHealth app either while they are an inpatient post-transplant, or at their first post-transplant clinic visit. Study personnel will assist participants assigned to the mHealth intervention arm with downloading the application and explain its functioning. Participants will then use the application to aid in immunosuppressant medication adherence post-transplant.
  Interventions: Other: mHealth Intervention

INTERVENTIONS:
Other: mHealth Intervention — The mHealth application will allow liver transplant recipients to see their medication regimen, record a video of themselves taking every dose, report side effects or symptoms, visualize their treatment progress, and access educational content. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review.
  Arms: mHealth Intervention

SUMMARY:
The investigators are interested in whether or not the use of a mobile health (mHealth) application increases the rate of immunosuppressant medication adherence among adult liver transplant recipients. The investigators aim to test this by randomly assigning transplant recipients to the intervention (use of an mHealth app to manage and track their immunosuppression regimen) or control arm (standard of care) upon discharge from their initial transplant hospitalization, and tracking medication adherence over time. The study population will be approximately 50 adult liver transplant recipients at the Johns Hopkins Hospital.

DETAILED DESCRIPTION:
In adult transplant recipients, poor adherence to immunosuppressant medications carries the risk of graft rejection, post-transplant complications, and increased healthcare costs. In adult liver transplant recipients, adherence to immunosuppressant drugs, as well as to general medical indications (e.g. avoiding alcohol intake), is imperative to short- and long-term outcomes. The rate of non-adherence to immunosuppressant medications in this population varies vastly, with reports ranging from 15-40%. Because of lacking objective and accurate non-adherence measurements, the true implications and prevalence of non-adherence is not yet well understood. Therefore, the investigators believe that mobile health (mHealth) technology has the potential to allow clinicians and researchers to more comprehensively address and understand non-adherence in adult liver transplant recipients. Additionally, an mHealth application with the ability to track symptoms, side effects, and alcohol cravings could provide clinicians with valuable information on post-transplant care.

We will use a mobile health platform that enables users to track dose-by-dose medication adherence through asynchronous, video directly observed therapy (DOT). This helps patients take their medication as prescribed and gives providers the assurance that their patients are supported and successful in treatment. DOT is the practice of watching a patient take every dose of medicine in-person, and has typically only been done in extreme cases because it can be both costly and burdensome: DOT is the standard of care for Tuberculosis treatment and has proven high-adherence rates. Through mHealth technology, DOT can be used more broadly and without added burden; emocha's technology allows this through enabling patients to use their mobile application to view their regimen, record themselves taking every dose of their medication, report side effects or symptoms, visualize their treatment progress, and access educational content. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review. The aim of this study is to conduct a randomized control trial to compare medication adherence between patients who use the mHealth application against controls who do not.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 22 years of age
* Receive a liver transplant at Johns Hopkins Hospital

Exclusion Criteria:

* Non-English speaking liver transplant recipients

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
12-week immunosuppression medication adherence | 12 weeks
  After 12 weeks in the study, patients will complete the 4-item immunosuppressant therapy adherence instrument (ITAS) to determine self-reported medication adherence (scores range from 0-12 with 0 indicating very poor adherence and 12 indicating perfect adherence). Additionally, immunosuppression level trends will be tracked via electronic medical record review to determine medication adherence.

SECONDARY OUTCOMES:
Feasibility of using the mHealth Application as Assessed by a Semi-Structured Interview and a 17-Item Survey | 12 weeks
  After 12 weeks in the study, participants will be asked to participate in a semi-structured phone interview in which they will answer questions regarding their medication adherence habits and their thoughts on how our mHealth technology was or was not helpful. They will also complete a 17-question post-satisfaction survey assessing their satisfaction levels with the mhealth technology. Responses in the 17-item survey are on a 7-item Likert scale, ranging from Strongly Agree to Strongly Disagree.
Alcohol Craving Assessment | 12 weeks
  As abstaining from alcohol is important following liver transplantation, we will administer a daily question through the mDOT app asking about alcohol craving and use. Patients who screen positive for alcohol craving and or use through the daily in-app question will be referred to a transplant social worker who will administer the Alcohol Craving Questionnaire Short Form.

CONTACTS AND LOCATIONS:
Overall Officials: Macey Henderson, JD, PhD, Principal Investigator — Johns Hopkins University; Andrew Cameron, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mor E, Gonwa TA, Husberg BS, Goldstein RM, Klintmalm GB. Late-onset acute rejection in orthotopic liver transplantation--associated risk factors and outcome. Transplantation. 1992 Nov;54(5):821-4. doi: 10.1097/00007890-199211000-00010. PMID 1279849
- [Background] O'Carroll RE, McGregor LM, Swanson V, Masterton G, Hayes PC. Adherence to medication after liver transplantation in Scotland: a pilot study. Liver Transpl. 2006 Dec;12(12):1862-8. doi: 10.1002/lt.20828. PMID 16773637
- [Background] Stilley CS, DiMartini AF, de Vera ME, Flynn WB, King J, Sereika S, Tarter RE, Dew MA, Rathnamala G. Individual and environmental correlates and predictors of early adherence and outcomes after liver transplantation. Prog Transplant. 2010 Mar;20(1):58-66; quiz 67. doi: 10.1177/152692481002000110. PMID 20397348
- [Background] Pinsky BW, Takemoto SK, Lentine KL, Burroughs TE, Schnitzler MA, Salvalaggio PR. Transplant outcomes and economic costs associated with patient noncompliance to immunosuppression. Am J Transplant. 2009 Nov;9(11):2597-606. doi: 10.1111/j.1600-6143.2009.02798.x. PMID 19843035
- [Background] Burra P, Germani G, Gnoato F, Lazzaro S, Russo FP, Cillo U, Senzolo M. Adherence in liver transplant recipients. Liver Transpl. 2011 Jul;17(7):760-70. doi: 10.1002/lt.22294. PMID 21384527
- [Background] Laederach-Hofmann K, Bunzel B. Noncompliance in organ transplant recipients: a literature review. Gen Hosp Psychiatry. 2000 Nov-Dec;22(6):412-24. doi: 10.1016/s0163-8343(00)00098-0. PMID 11072057
- [Background] Hathaway DK, Combs C, De Geest S, Stergachis A, Moore LW. Patient compliance in transplantation: a report on the perceptions of transplant clinicians. Transplant Proc. 1999 Jun;31(4A):10S-13S. doi: 10.1016/s0041-1345(99)00113-x. No abstract available. PMID 10372033
- [Background] Dobbels F, Vanhaecke J, Desmyttere A, Dupont L, Nevens F, De Geest S. Prevalence and correlates of self-reported pretransplant nonadherence with medication in heart, liver, and lung transplant candidates. Transplantation. 2005 Jun 15;79(11):1588-95. doi: 10.1097/01.tp.0000158430.06507.87. PMID 15940050
- [Background] Nahid P, Dorman SE, Alipanah N, Barry PM, Brozek JL, Cattamanchi A, Chaisson LH, Chaisson RE, Daley CL, Grzemska M, Higashi JM, Ho CS, Hopewell PC, Keshavjee SA, Lienhardt C, Menzies R, Merrifield C, Narita M, O'Brien R, Peloquin CA, Raftery A, Saukkonen J, Schaaf HS, Sotgiu G, Starke JR, Migliori GB, Vernon A. Executive Summary: Official American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America Clinical Practice Guidelines: Treatment of Drug-Susceptible Tuberculosis. Clin Infect Dis. 2016 Oct 1;63(7):853-67. doi: 10.1093/cid/ciw566. PMID 27621353
- [Background] Chisholm MA, Lance CE, Williamson GM, Mulloy LL. Development and validation of the immunosuppressant therapy adherence instrument (ITAS). Patient Educ Couns. 2005 Oct;59(1):13-20. doi: 10.1016/j.pec.2004.09.003. PMID 16198214
- [Background] Singleton, E.G., Tiffany, S.T. & Henningfield, J.E. (2000). Alcohol Craving Questionnaire (ACQ-NOW): Background, Scoring, and Administration (Manual). Baltimore, MD: Intramural Research Program, National Institute on Drug Abuse.
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829